CLINICAL TRIAL: NCT04839770
Title: The Minimally Invasive Endoscopic Surgery With the Axonpen System for Spontaneous Intracerebral Hemorrhage (MIECH): An Open-label, Non-randomized, Single-arm Pilot Study
Brief Title: MIECH: The Minimally Invasive Endoscopic Surgery With the Axonpen System for Spontaneous Intracerebral Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clearmind Biomedical Inc. (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MIECH-2020-01
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Intracerebral Hemorrhage; Cerebral Hemorrhage; Intracranial Hemorrhage; Basal Ganglia Hemorrhage
Keywords: Intracerebral Hemorrhage; Cerebral Hemorrhage; Intracranial Hemorrhage; ICH; Stroke; Endoscopic Hematoma Evacuation; Minimally Invasive Surgery; Endoscopic Neurosurgery
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Basal Ganglia Hemorrhage; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axonpen (Experimental): Subjects will receive minimally invasive endoscopic surgery using the Axonpen™ system for early hematoma evacuation (within 48 hours post-ictus).
  Interventions: Device: Axonpen system

INTERVENTIONS:
Device: Axonpen system — The Axonpen™ system, containing the Axonpen and the Axonmonitor, has been cleared for the illumination and visualization of intracranial tissue and fluids and the controlled aspiration of tissue and/or fluid during surgery of the ventricular system or cerebrum.
  The Axonpen is a neuroendoscope integrated with suction (sourced from hospital vacuum) and irrigation (sourced from third-party saline infusion bag) functions. The Axonmonitor is used for view and storage of the endoscopic image. The Axonpen™ system is intended to optimize the procedure of minimally invasive neurosurgery for early ICH evacuation.

SUMMARY:
The primary objective of this trial is to provide preliminary safety data of minimally invasive endoscopic surgery using the Axonpen™ system for spontaneous intracerebral hemorrhage (ICH). The effectiveness of the Axonpen™ system in early hematoma removal and the surgical impact on subject's functional recovery will also be evaluated.

The Axonpen™ system, consisting of a neuroendoscope (Axonpen) and a monitor (Axonmonitor), is cleared by FDA and indicated for the illumination and visualization of intracranial tissue and fluids and the controlled aspiration of tissue and/or fluid during surgery of the ventricular system or cerebrum.

DETAILED DESCRIPTION:
In the present trial, the FDA-cleared Axonpen™ system was applied on the ICH surgery. The Axonpen™ System is a neuroendoscope combined with the functions of hematoma aspiration and irrigation, aiming to minimize surgical brain injury, optimize surgical procedure, and be available for early hematoma evacuation.

The technique of minimally invasive endoscopic neurosurgery for ICH is still considered in development; however, a retrospective study [Kuo et al.] has shown that early and complete evacuation of ICH may lead to improved outcomes in selected patients, where the neurosurgeons utilized combination of the existing instruments, such as a rod-lens endoscope with irrigation system and a suction coagulator, to enable visualization, aspiration, and irrigation of the hematoma to be worked simultaneously. The technology employed and the results revealed in the previous study provide a proof of concept for the Axonpen™ system, and also imply that the current device could be safe and effective in the management of ICH.

ELIGIBILITY:
Inclusion Criteria:

Patients who fulfill ALL the inclusion criteria will be enrolled:

1. Age 20-80 years, all genders/sexes are inclusive;
2. Evidence of a spontaneous basal ganglia ICH on CT scan;
3. Patient, or a family member with legally authorized responsibility, has given informed consent;
4. GCS of 6-14;
5. Volume of hematoma in range of 30-80 ml as measured by the ABC/2 method;
6. Can receive surgical treatment within 48 hours after ictus.

Exclusion Criteria:

Patients who fulfill ANY ONE of the exclusion criteria should not be enrolled:

1. Previous symptomatic stroke with neurological sequelae (per history or as seen on initial CT scan);
2. ICH known or suspected by study investigator to be secondary to aneurysm, vascular malformation, hemorrhagic transformation of ischemic stroke, cerebral venous thrombosis, thrombolytic therapy, tumor, or infection;
3. Acute or active infection signs requiring treatment at the time of admission;
4. Significant ventricular extension of the hemorrhage; more than 30 mL of intraventricular hemorrhage;
5. Refractory elevated ICP after placement of an EVD (external ventricular drain);
6. Severe pre-existing physical or mental disability or severe co-morbidity which might interfere with assessment of outcome;
7. Minimally invasive neurosurgery could not be commenced within 48 hours of onset. The case shall be excluded when the time of onset cannot be estimated and is judged with controversy by the investigator;
8. The hematological effects of any previous anticoagulants are not completely reversed (platelet count < 100 × 10^3/μL; international normalized ratio (INR) > 1.4);
9. Hereditary or acquired hemorrhagic diathesis or coagulation factor deficiency;
10. Any condition that could impose hazards to the patient with the MIN or affect the participation of the patient in the study. The judgment is left to the discretion of the investigator;
11. Major surgery within the preceding 14 days which poses risk in the opinion of the investigator;
12. Any history or current evidence suggestive of venous or arterial thrombotic events within the previous 12 months, including clinical, ECG, laboratory, or imaging findings;
13. Use of heparin, low-molecular weight heparin, GPIIb/IIIa antagonist, antiplatelet agents, or oral anticoagulation (e.g., warfarin, factor Xa inhibitor, thrombin inhibitor) within the previous 14 days, irrespective of laboratory values;
14. Pregnancy, breast-feeding, or positive pregnancy test (either serum or urine) (Woman of child-bearing potential must have a negative pregnancy test prior to the study procedure.);
15. Participation in any investigational study in the last 30 days;
16. Known terminal illness or planned withdrawal of care or comfort care measures.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of Mortality | 30 days
  Safety will be assessed by determining mortality within 30 days post-operation for all subjects
Number of Adverse events (AEs), Serious Adverse Events (SAEs), and Unanticipated Device Effects (UDEs) | 180 days
  AEs, SAEs, and UDEs will be observed from the beginning of the surgery until the last follow-up visit (Day 180) for safety monitoring, and their relation to the study device will be analyzed

SECONDARY OUTCOMES:
Hemorrhage volume | 6 and 72 hours
  Residual hematoma will be measured via 6 & 72 hours post-operation CT. Reduction (%) of hemorrhage volume will be assessed by comparing with pre-operation CT
Glasgow Coma Scale (GCS) | 180 days
  Clinical assessment for level of consciousness and responsiveness before and after surgery (Assessed by the sum of E/V/M scores. E: Eye opening, 1 = None - 4 = Spontaneous. V: Verbal response, 1 = None - 5 = Normal conversation. M: Motor response, 1 = None - 6 = Normal)
modified Rankin Scale (mRS) | 180 days
  Functional outcomes will be measured via mRS at 72 hours and 7 days post-operation, hospital discharge, and 40, 90, 180 days follow-up visits (Scale ranges from 1 to 7, 1 = No symptoms - 7 = Dead)
Glasgow Outcome Scale Extended (GOSE) | 180 days
  Functional outcomes will be measured via GOSE at 72 hours and 7 days post-operation, hospital discharge, and 40, 90, 180 days follow-up visits (Scale ranges from 1 to 8, 1 = Death - 8 = Upper good recovery)
Length of ICU | Number of days from admission, up to 180 days
  Duration of stay in the ICU
Length of hospitalization | Number of days from admission to discharge, up to 180 days
  Duration of stay in the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital (Linkou Branch), Taoyuan District, Taiwan

REFERENCES:
- [Background] Kuo LT, Chen CM, Li CH, Tsai JC, Chiu HC, Liu LC, Tu YK, Huang AP. Early endoscope-assisted hematoma evacuation in patients with supratentorial intracerebral hemorrhage: case selection, surgical technique, and long-term results. Neurosurg Focus. 2011 Apr;30(4):E9. doi: 10.3171/2011.2.FOCUS10313. PMID 21456936